CLINICAL TRIAL: NCT07215546
Title: Enhanced Sternal Closure With Montage or Montage-CT to Evaluate Post-Operative Opioid Use Following Median Sternotomy
Status: Enrolling by invitation | Type: Observational
Sponsor: Abyrx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Abyrx PMRCT 25-002
Record Dates: First submitted 2025-09-25; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Retrospective Review; Cerclage; Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Control: Standard sternal cerclage closure with no settable putty applied in the timeframe (less than one year) immediately preceding use of the test device or concurrently.
- Montage or Montage CT: Standard sternal cerclage closure (typically a minimum of 6 single loop closures) with application of Montage or Montage-CT Settable Resorbable Bone Putty to the cut sternal edge at the time of closure.
  Interventions: Device: Montage or Montage CT

INTERVENTIONS:
Device: Montage or Montage CT — Application of Montage or Montage-CT Settable Resorbable Bone Putty to the cut sternal edge at the time of closure.
  Groups: Montage or Montage CT

SUMMARY:
This is a retrospective study based on analysis real world data obtained from hospitals that have adopted use of Montage or Montage-CT for use following sternotomy. The analysis will report the post-operative use of analgesic medication (including opioids) and compare the use against a control group consisting of patients operated by the same surgeon concurrently or prior to adoption of Montage or Montage-CT for use in sternotomy closure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 19 years of age.
2. Underwent non-emergent cardiac surgery (isolated coronary artery by-pass grafting and/or isolated valve surgery).
3. Full median sternotomy approach - with/without cardiopulmonary bypass.

Exclusion Criteria:

1. Recent CPR.
2. Previous cardiac surgery (redo sternotomy).
3. Emergency surgery (operative intervention within 24 hrs of assessment).
4. Chronic lung disease.
5. BMI > 40.
6. Use of sternal plate systems for closure.
7. Recent antiplatelet therapy.
8. Previous radiotherapy to the chest; receiving immunosuppressive therapy or have a current immunosuppressive condition.
9. Active systemic infection (.i.e: endocarditis).
10. Cognitive impairment (confusion, dementia, Alzheimers, current substance abuse).
11. History of malignancies within past year (except squamous or basal cell carcinoma of the skin that has been treated; no recurrence)
12. Recent history of drug or alcohol abuse.
13. Females who are pregnant, nursing or of childbearing potential who are not practicing a birth control method with high reliability.
14. Postsurgical life expectancy < 90 days in the opinion of the investigator.

14. Moderate or severe pectus deformity. 16. Participation in another clinical trial. 17. Patients who had Patient-Controlled Analgesia (PCA) devices after surgery. 18. Patients who received a local anesthetic treatment and/or device on the sternum intraoperatively during surgery (e.g. On-Q Pain Relief System, Exparel etc)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females age > 19 years of age who have undergone non-emergent cardiac surgery (coronary artery by-pass grafting [CABG] and/or single valve replacement procedure).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Cumulative Opiod Dose | From admission until end of treatment/discharge, up to 8 weeks
  1. Cumulative opioid dose (COD) is measured from entry into the postoperative ICU through the time of achieving hospital discharge criteria. Opioid use will be quantified in morphine equivalents, using conversion factors based on Von Korff, et al.

SECONDARY OUTCOMES:
Time to Discharge | From admission until end of treatment/discharge, up to 8 weeks
  Postoperative time to achieving hospital discharge criteria (TTHDC) measured in hours from entry into the postoperative ICU to the time a patient meets hospital discharge criteria.
Time to Opioid Cessation | From admission until end of treatment/discharge, up to 8 weeks
  Time to opioid cessation (TTOC) measured in hours from entry into the postoperative ICU to the first time point at which a patient achieved a sustained period of at least 24 consecutive hours.
Percent Discharged with Opioid Prescription | From admission until end of treatment/discharge, up to 8 weeks
  Percentage of patients discharged with an opioid prescription (DWOP) based on the number of patients who received a prescription for an opioid medication at hospital discharge.
Percent without Opioid Use | From admission until end of treatment/discharge, up to 8 weeks
  Percentage of patients with no opioid analgesic use (NOU) based on the number of patients who did not receive any opioid medication from entry into the postoperative ICU through the time of achieving hospital discharge criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Aniq Darr, Ph.D., Study Director — Abyrx, Inc.
Locations (2):
- United States (2):
  - NCH Rooney Heart Institute, Naples, Florida
  - Washington University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Losanoff JE, Richman BW, Jones JW. Risk analysis of deep sternal wound infection and mediastinitis in cardiac surgery. Thorac Cardiovasc Surg. 2002 Dec;50(6):385. doi: 10.1055/s-2002-35738. No abstract available. PMID 12457323
- [Background] Meyerson J, Thelin S, Gordh T, Karlsten R. The incidence of chronic post-sternotomy pain after cardiac surgery--a prospective study. Acta Anaesthesiol Scand. 2001 Sep;45(8):940-4. doi: 10.1034/j.1399-6576.2001.450804.x. PMID 11576043
- [Background] Kalso E, Mennander S, Tasmuth T, Nilsson E. Chronic post-sternotomy pain. Acta Anaesthesiol Scand. 2001 Sep;45(8):935-9. doi: 10.1034/j.1399-6576.2001.450803.x. PMID 11576042
- [Background] Ingason AB, Geirsson A, Gudbjartsson T, Muehlschlegel JD, Sigurdsson MI. The Incidence of New Persistent Opioid Use Following Cardiac Surgery via Sternotomy. Ann Thorac Surg. 2022 Jan;113(1):33-40. doi: 10.1016/j.athoracsur.2021.04.030. Epub 2021 Apr 27. PMID 33930358
- [Background] Brown CR, Chen Z, Khurshan F, Groeneveld PW, Desai ND. Development of Persistent Opioid Use After Cardiac Surgery. JAMA Cardiol. 2020 Aug 1;5(8):889-896. doi: 10.1001/jamacardio.2020.1445. PMID 32584934
- [Background] Li AE, Fishman EK. Evaluation of complications after sternotomy using single- and multidetector CT with three-dimensional volume rendering. AJR Am J Roentgenol. 2003 Oct;181(4):1065-70. doi: 10.2214/ajr.181.4.1811065. No abstract available. PMID 14500232
- [Background] Losanoff JE, Jones JW, Richman BW. Primary closure of median sternotomy: techniques and principles. Cardiovasc Surg. 2002 Apr;10(2):102-10. doi: 10.1016/s0967-2109(01)00128-4. PMID 11888737
- [Background] McGregor WE, Trumble DR, Magovern JA. Mechanical analysis of midline sternotomy wound closure. J Thorac Cardiovasc Surg. 1999 Jun;117(6):1144-50. doi: 10.1016/s0022-5223(99)70251-5. PMID 10343263
- [Background] Lemaignen A, Birgand G, Ghodhbane W, Alkhoder S, Lolom I, Belorgey S, Lescure FX, Armand-Lefevre L, Raffoul R, Dilly MP, Nataf P, Lucet JC. Sternal wound infection after cardiac surgery: incidence and risk factors according to clinical presentation. Clin Microbiol Infect. 2015 Jul;21(7):674.e11-8. doi: 10.1016/j.cmi.2015.03.025. Epub 2015 Apr 14. PMID 25882356